CLINICAL TRIAL: NCT01067001
Title: Open Label, Balanced, Randomized, Two-treatment, Two-sequence, Two-period, Single-dose, Crossover, Bioequivalence Study in Normal, Healthy, Adult, Human Subjects Under Fasting Condition.
Brief Title: Minocycline HCl Extended Release Tablets 135 mg Oral Bioequivalence Study
Acronym: Minocycline
Status: Completed | Type: Observational
Sponsor: Amneal Pharmaceuticals Co. India Private Limited (Industry)
Responsible Party: Dr. Nikunj Patel, Amneal Pharmaceuticals Co. India Private Limited
Other Study IDs: Amneal-10-01
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 2 Way Crossover: 2 Way Crossover bioequivalence study
- Subjects will be randomly divided in to 2 groups.: A total of 18 normal, healthy, adult, human subjects will be enrolled in the study.

SUMMARY:
To determine single-dose oral bioequivalence of Minocycline HCl Extended Release Tablets 135 mg manufactured by Amneal Pharmaceuticals Co.(I)Pvt. Ltd., India and SOLODYN® (minocycline hydrochloride) Extended Release Tablets 135 mg Manufactured for Medicis, The Dermatology Company, Scottsdale, AZ 85256, by Wellspring Pharmaceutical Canada Corp., Oakville, Ontario L6H 1M5 in normal, healthy, adult, human subjects under fasting condition.

DETAILED DESCRIPTION:
Subjects will be fasted for at least 10 hours prior to scheduled time for dosing. As per the randomization schedule, one tablet of test or reference product will be administered to each subject with 240 mL of water at ambient temperature in each period.

Twenty four samples will be collected from each subject during each period. The venous blood samples (5 mL each) will be withdrawn at pre-dose (before dosing, in the morning of the day of dosing) and at 1.00, 2.00, 2.50, 3.00, 3.25, 3.50, 3.75, 4.00, 4.25, 4.50, 5.00, 5.50, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 48.00, 72.00, 96.00, and 120.00 hours after dosing. The samples collected at 48.00, 72.00, 96.00, and 120.00 hours after dosing will be on an ambulatory basis (i.e. on separate visit).

After collecting the blood samples from all the subjects at each sampling time point, samples will be centrifuged under refrigeration with machine set at 3000 rpm, 10 minutes and 4oC. After centrifugation, the plasma samples will be separated and transferred into respective prelabeled polypropylene tubes. These polypropylene tubes will be stored below -20°C for a maximum period of 12 hours and then they will be stored at -70°C ± 20°C until withdrawn for analysis.

Samples from all the subjects completing both periods of the study as per the approved protocol will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

Healthy human subjects aged between 18 and 45 years.(including both) Subjects with a BMI between 18.5 - 24.9 Kg/m2 (including both) and body weight not less than 45 Kgs.

Subjects with normal health as determined by personal medical history, clinical examination, and laboratory examinations including serological tests Subjects having normal 12-lead electrocardiogram (ECG). Subjects having normal chest X-Ray (P/A view). Subjects able to communicate effectively. Subjects willing to give written informed consent and adhere to all the requirements of this protocol.

Female subjects who are postmenopausal or surgically sterile. Female subjects practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD) or abstinence.

Exclusion Criteria:

* Subjects having contraindications or hypersensitivity to minocycline or related group of drugs.
* History or presence of any medical condition or disease according to the opinion of the physician.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
* History or presence of significant alcoholism or drug abuse in the past one year.
* History or presence of significant smoking (more than 10 cigarettes or bidis/day or consumption of tobacco products).
* Difficulty with donating blood.
* Difficulty in swallowing solids like tablets or capsules.
* Systolic blood pressure less than 90 mm Hg or more than 140 mm Hg.
* Diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
* Pulse rate less than 50 beats/minute or more than 100 beats/minute.
* Use of any prescribed medication during last two weeks or OTC medicinal products during the last one week preceding the first dosing.
* Major illness during 3 months before screening.
* Participation in a drug research study within past 3 months.
* Donation of blood in the past 3 months before screening.
* Female subjects demonstrating a positive pregnancy screen.
* Female subjects who are currently breast-feeding.
* Female subjects with child bearing potential using prohibited contraceptive method (Oral, Injectable or Implantable hormonal agents).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 18 normal, healthy, adult, human subjects will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The following parameters will be considered as primary end points to determine the bioequivalence of test and reference products: Cmax, AUC0-t and AUC0-INF

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nikunj Patel, MD, Pharmacology, Study Director — Director, CRO
Locations (1):
- Hyderabad, Andharapradesh, India